CLINICAL TRIAL: NCT04497051
Title: Using CT-DSA With Deformable Registration Technique to Predict Efficacy in Preoperative Embolization for Spinal Metastasis
Brief Title: CT-DSA Evaluation of Embolization in Debulking Spinal Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001028RINB
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-03

CONDITIONS: Spinal Metastases; Surgery
Keywords: vertebra; embolization; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embolized patients: subjects receiving preoperative embolization for aggressive spinal debulking surgery
  Interventions: Diagnostic Test: CT-DSA

INTERVENTIONS:
Diagnostic Test: CT-DSA — CTA before and after embolization

SUMMARY:
Vertebra is one of the most common site of metastatic disease, which may cause severe pain or neurological deficit. Decompressive surgery or radiation therapy are of limited efficacy and recurrence is very likely. Debulking surgery usually has better local control and survival benefit. However, debulking surgery often accompany with massive blood loss, which may cause hemorrhagic shock or death. It is known that intraoperative blood loss is associated with tumoral vascularity. However, there is current no objective method to evaluate vascularity status. On the other hand, preoperative embolization is considered as major method to decrease blood loss. There is also objective method to evaluate the embolization effect. By our innovative dual energy computed tomography angiography - digital subtraction angiography (CT-DSA), the tumoral vascularity status and embolization effect of spinal tumor can be objectively assessed. We aim to utilize CT-DSA to investigate spinal tumor, in a hope to find out correlation of vascularity status, embolization method, and surgical outcome, which can help individual disease status and tailored treatment decision.

Key word: spine/embolization/computed tomography

DETAILED DESCRIPTION:
Vertebral osseus metastasis, can cause neoplastic spinal cord compression and neurological deficit. The treatment strategy depend on the pathological type, performance status, and life expectancy. The goal of treatment is to avoid neurological deterioration, to keep functional life, and to control bone pain. Treatment strategy involve multidisciplinary approaches between spinal surgeon, medical and radiation oncologist, and radiologist. When presence of acute neurological deterioration or intractable pain due to neoplastic compression or vertebral instability, surgical approach is often warranted. In term of surgical approach, simple decompression and fixation is often applied, but the long-term control rate is suboptimal. Aggressive spinal surgery, including extensive debulking surgery or spondylectomy, has relative longstanding effect to maintain neurological and oncological outcome.

Despite relative good outcome of aggressive spinal surgery, it is a relative massive procedure in which life-threatening blood loss commonly occur. To achieve better surgical outcome and decrease complication, preoperative embolization is suggested to control blood loss . The procedure is performed by an interventional radiologist to deliver embolic agent into vascular pedicles of target vertebra, in hope to achieve optimal devascularization of the tumour. The concept is simple and the similar procedure has been performed thousands of times in the world. However, its efficacy and utilization are not yet proven by clinical trials. When and how to perform this procedure largely depends on experience of operating interventional radiologist.

CT is an important imaging tool for spinal disease. Because of its rapid acquisition, adequate resolution, and easy reformatting, it is optimal for intolerable patients. Nevertheless, osseous structure is extremely radiopaque, evaluation of tumoral enhancement in vertebrae is not easy. Nevertheless, the enhancement of osseous tumour can be evaluated with advanced subtraction reformatting technique. The technique is similar to digital subtraction angiography (DSA) of catheter angiography, and we call it CT-DSA image. As compared with traditional catheter-based DSA, CT-DSA has following additional advantages: 1) non-invasiveness; 2) non-selective enhancement of the target; 3) allowing multiplanar reformatting and additional post-processing and quantification. The tool is very versatile to investigate the vascularity of the vertebral neoplasm. In our earlier result, we found the CT-DSA has good correlation with DSA in vascularity assessment, suggestive of its utilization in pre-operative and pre-embolization evaluation of spinal tumour. It can be used in semi-quntitative and quantitative fashion.

Traditionally, the efficacy of embolization is determined by surgical outcome, usually with gold standard of blood loss. However, blood loss is determined by many different factors, including tumor volume, surgical technique, and other anatomical factors. Using CT-DSA, evaluation of the embolization effect directly is possible. As the study can be repeated after embolization, the interval change can be observed with objective measurement.

In summary, using CT-DSA, it is possible to evaluate the vascularity of the osseous tumour and efficacy of devascularization after embolization before surgery. We can therefore design study to test efficacy of different intervention strategy, and find out the more beneficial indication, which can incorporate into clinical workflow and help patients.

Purpose

1. The establish subjective risk classification of debulking surgery in term of tumour vascularity
2. To subjectively evaluate efficacy of preoperative embolization
3. To design appropriate clinical workflow in management of patient with vertebral malignancy

Importance Vertebrae is 3rd most common site of metastatic malignancy, and is usually warrant aggressive spinal surgery. Since preoperative embolization is commonly done in this patient, it needs subjective tool to assess its efficacy and clear indication. By using CT-DSA, there is potential to provide tailored strategy of patient management before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with clinical diagnosis for thoracolumbar vertebral primary or metastatic malignancy
2. Eligible for aggressive spinal surgery, including debulking and en bloc spondylectomy
3. Life expectancy more than 6 months
4. Serum creatinine less than 1.5 mg/dL

Exclusion Criteria:

1. Age less than 20 year old
2. Woman in pregnancy or breast feeding
3. Serious allergic reaction to contrast medium
4. Instable neurological condition warrant urgent operation

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with clinical diagnosis for thoracolumbar vertebral malignancy who can receive preoperative emoblization
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
estimated blood loss during surgery | 24 hours
  blood lose in debulking spinal surgery

SECONDARY OUTCOMES:
transfusion amount | 24 hours
  perioperative blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Heng Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan